CLINICAL TRIAL: NCT02918669
Title: Study to Investigate the Long Term Survivorship of Coflex CT Study: Sub-Analysis of 24 Month Spinous Process Fractures Via Post-60 Month CT Scan
Brief Title: Study to Investigate the Long Term Survivorship of Coflex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paradigm Spine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PAS001a
Record Dates: First submitted 2016-04-27; First posted 2016-09-29 (Estimated); Results first posted 2019-07-08 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Spinal Fractures
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- coflex (Experimental): Patients who received the coflex Device in the IDE Study and presented with a spinous process fracture at 24 months (identified by independent radiographic review lab). Patients will undergo a CT Scan.
  Interventions: Radiation: CT Scan

INTERVENTIONS:
Radiation: CT Scan — Patients in the coflex IDE Study who presented at 24 months with a spinous process fracture that will undergo a CT Scan to evaluate the evidence or healing of fracture post-60 months.
  There are no other interventions. It is just a onetime CT post 60 month time point.

SUMMARY:
Examine the long-term survivorship via CT Scan of the coflex in patients who presented with spinous process fracture(s) at 24 months in the Paradigm Spine coflex IDE Study.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm, radiographic evaluation of all coflex IDE patients who presented with a spinous process fracture at 24 months as identified by independent radiographic review (using X-ray or CT). All patients were enrolled and followed through 60 months under the IDE and extended follow-up protocol.

The specific objective of this CT Study is to perform a sub-analysis of the patients with 24 month spinous process fracture(s) via a CT scan at post-60 months. A CT Scan will be performed and analyzed by an independent radiographic review lab for evidence of fracture or healing at the long term timepoint.

ELIGIBILITY:
Inclusion Criteria:

* Participant in coflex IDE Study
* Willing and able to give informed consent
* Spinous process fracture identified by site and/or radiographic lab at 24 months

Exclusion Criteria:

* Subjects who died, were withdrawn or withdrew consent to participate in the study
* Subjects who are pregnant, or planning to become pregnant, during the course of this study
* Subjects who have cancer, whether active or in remission

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2017-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hal Mathews, MD, Study Director — Paradigm Spine

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Coflex: Patients who received the coflex Device in the IDE Study and presented with a spinous process fracture at 24 months (identified by independent radiographic review lab). Patients will undergo a CT Scan.
  CT Scan: Patients in the coflex IDE Study who presented at 24 months with a spinous process fracture that will undergo a CT Scan to evaluate the evidence or healing of fracture post-60 months.
  There are no other interventions. It is just a onetime CT post 60 month time point.
Period: Overall Study
Arm/Group | Coflex
Started | 12
Completed | 8
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Patients who presented with spinous process fractures at 24 months in the Paradigm Spine coflex® IDE Study.
Arm/Group | Coflex
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
CT Scan of the coflex® in patients who presented with spinous process fractures at 24 months [Count of Participants; unit: Participants] | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Radiographic Analysis of Evidence of Fracture or Healing Based on CT Scan
Description: Any coflex patients with radiographic observations of spinous process fracture at post-24 months, will be examined via CT at 5 years for evidence of fracture or of healing.
Time Frame: Post-60 Months
Population: To examine the long-term survivorship via CT Scan of the coflex in patients who presented with spinous process fractures at 24 months in the Paradigm Spine coflex IDE Study.
Measure: Count of Participants; unit: Participants
Arm/Group | Coflex
Number analyzed (Participants) | 8
Participants | 8

2. Post Hoc Outcome: Fracture Location
Description: 0 None; no evidence of spinous process fracture
  1. Posterior avulsion; presence of a fracture pattern consistent with lumbar spinous process avulsion fractures
  2. Posterior to implant wings; presence of a spinous process fracture posterior
  3. Coincident with implant wings: presence of a spinous process fracture in the same coronal plane as the implant wings
  4. Anterior to implant wings; presence of a spinous process fracture anterior to the implant wings
  5. Indeterminate; assessment cannot be made due to technical factors such as obscured anatomy due to the device wings, poor contrast, high parallax or significant artifacts that result in images being of non-diagnostic quality
Time Frame: >/= 5 years
Measure: Number; unit: fractures
Arm/Group | Coflex
Number analyzed (Participants) | 8
fractures
  Anterior to wings | 6
  Coincident with implant wings | 2

3. Post Hoc Outcome: Fracture Displacement
Description: 0 N/A; no spinous process fracture reported
  1. Non-displaced; no evidence of a displaced spinous process fracture
  2. Displaced; presence of a displaced spinous process fracture. No contact between the fragment and the remaining vertebra should exist, and at least 2 mm wide gap should exist at a point along the fracture gap
  3. Indeterminate; assessment cannot be made due to technical factors such as obscured anatomy due to the device wings, poor contrast, high parallax or significant artifacts that result in images being of non-diagnostic quality
Time Frame: >/= 5 years
Measure: Number; unit: fractures
Arm/Group | Coflex
Number analyzed (Participants) | 8
fractures
  Displaced | 5
  Non-Displaced | 6

4. Post Hoc Outcome: Fracture Healing
Description: 0 N/A; no spinous process fracture reported
  1. Not healed; no evidence of a spinous process fracture healing
  2. Healed; presence of a healed spinous process fracture
  3. Remodeled; fracture line is absent due to bone remodeling at the site of a previously detected fracture
  4. Indeterminate - no follow-up imaging available; no images are available at time points later than the time point when the fracture was identified
  5. Indeterminate - inadequate image quality; the quality of available images is inadequate to determine the fracture healing status
  6. Indeterminate - implant obscures fracture; the coflex implant obscures visualization of the fracture line so healing cannot be determined
Time Frame: >/= 5 years
Measure: Number; unit: fractures
Arm/Group | Coflex
Number analyzed (Participants) | 8
fractures
  Healed | 4
  Remodeled | 3
  Not Healed | 2
  Indeterminate | 2

ADVERSE EVENTS:
Description: Adverse events were not monitored/assessed as part of this study. The only data collected was the CT scan which was reviewed by an independent radiographic lab.
Groups:
- Coflex: Patients in the coflex IDE Study who presented at 24 months with a spinous process fracture that will undergo a CT Scan to evaluate the evidence or healing of fracture post-60 months. There are no other interventions. It is just a onetime CT post 60 month time point.
Arm/Group | Coflex
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2016-05-02): https://cdn.clinicaltrials.gov/large-docs/69/NCT02918669/ICF_000.pdf
  • Study Protocol (2016-04-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT02918669/Prot_001.pdf